CLINICAL TRIAL: NCT06353659
Title: The Diagnostic Value of Contrast-enhanced Ultrasound in Acute Kidney Injury in Intensive Care Unit
Brief Title: The Diagnostic Value of Contrast-enhanced Ultrasound in Acute Kidney Injury in ICU
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Cui Ligang, Chief Physician, Peking University Third Hospital
Other Study IDs: M2024077
Record Dates: First submitted 2024-03-05; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Intensive Care Unit; Acute Kidney Injury; Ultrasound
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with acute kidney injury (AKI): Patient diagnosed with AKI according to kidney disease improving global outcomes (KDIGO) 2012 criteria
  Interventions: Diagnostic Test: Contrast-enhanced Ultrasound
- Patients without AKI: Patient diagnosed without AKI according to kidney disease improving global outcomes (KDIGO) 2012 criteria
  Interventions: Diagnostic Test: Contrast-enhanced Ultrasound

INTERVENTIONS:
Diagnostic Test: Contrast-enhanced Ultrasound — Patients with acute kidney injury high risk factors (KDIGO 2012) will undergo a contrast-enhanced ultrasound within 24 hours of admission to the ICU

SUMMARY:
The goal of this observational study is to quantitatively assess the renal microcirculation changes by contrast-enhanced ultrasound (CEUS) and to obtain systemic hemodynamic information by ultrasound Doppler at the same time, to analyze the relationship between renal microcirculation changes and systemic hemodynamic changes, and to explore the diagnostic value of CEUS in critically ill acute kidney injury.

DETAILED DESCRIPTION:
The main questions it aims to answer are:

1. To explore the quantitative parameters of contrast-enhanced ultrasound which can reflect the changes of renal microcirculation。
2. To explore the relationship between renal microcirculation and systemic hemodynamics。
3. To explore the value of quantitative evaluation of renal microcirculation changes by contrast-enhanced ultrasound in the diagnosis of acute kidney injury

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years old
* First admission to ICU < 24h after admission and expected ICU stay ≥48 hours
* Acute kidney injury risk factors (KDIGO 2012)
* Contrast-enhanced ultrasound

Exclusion Criteria:

* Known severe chronic kidney disease (CKD≥ stage 4) or undergoing hemodialysis treatment
* Kidney transplantation or renal malignancy
* Terminal stage of malignant tumor
* Pregnancy
* Renal artery stenosis or renal vein thrombosis
* The quality of CEUS images is poor, and quantitative analysis cannot be performed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Through literature review, the latest meta-analysis results showed that the area under the curve of CEUS parameters for diagnosing AKI was 0.84 and the width of the confidence interval was 0.22. When α=0.05, the sample size N=54 was obtained by PASS software. Considering the 10% shedding rate, 60 patients were expected to be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Acute kidney injury (according to KDIGO 2012 criteria) | Through study completion, an average of 7 days
  Acute kidney injury occur or not

CONTACTS AND LOCATIONS:
Overall Officials: Ligang Cui, Dr, Principal Investigator — Department of Ultrasound, Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: No